CLINICAL TRIAL: NCT03725345
Title: Genetic and Neural Factors in Alcohol-Related Cognition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: HM20013938; K01AA026647 (NIH)
Record Dates: First submitted 2018-10-29; First posted 2018-10-31 (Actual); Results first posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Alcohol Abuse
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alcohol Group (Active Comparator): Participants who have recently consumed alcohol.
  Interventions: Behavioral: MRI Scanner
- No Alcohol Group (Sham Comparator): Participants who have not recently consumed alcohol.
  Interventions: Behavioral: MRI Scanner

INTERVENTIONS:
Behavioral: MRI Scanner — Participants will enter the MRI scanner and complete a series of computer tasks that include noise blasts while undergoing brain scans that measure the structure and function of the brain

SUMMARY:
This study examines the genetic factors that impact cognitive processes and behavior after alcohol consumption. Participation in this project will contribute to a better understanding of cognitive factors that influence alcohol misuse.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* No current or regular use of prescribed or illicit psychoactive drugs
* Free of major health problems (e.g., diabetes, HIV, Parkinson's disease)
* Free of neurological or psychiatric disorders
* No current drug abuse (e.g., recreational drug use).
* Right-hand dominant
* Free of claustrophobia
* Free of pregnancy or suspected pregnancy
* Absent MRI risk factors (e.g., implanted medical device, body mass index > 35, braces)
* Free of medical conditions that render individuals with overly sensitive hearing
* Non-naive to alcohol consumption

Exclusion Criteria:

* Not meeting the inclusion criteria listed above

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2023-07-11 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Chester, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The results being reported apply only to Aim 4 of the grant. Aims 1-3 focused on analyzing existing archival genomic data and were covered by another protocol, which was not entered into CT.gov, as those aims did not meet the definition of a clinical trial and were approved under a different IRB protocol number and approval process than Aim 4.
Groups:
- Alcohol Group: Participants who have recently consumed alcohol. MRI Scanner: Participants will enter the MRI scanner and complete a series of computer tasks that include noise blasts while undergoing brain scans that measure the structure and function of the brain. The results being reported apply only to Aim 4 of the grant.
- No Alcohol Group: Participants who have not recently consumed alcohol. MRI Scanner: Participants will enter the MRI scanner and complete a series of computer tasks that include noise blasts while undergoing brain scans that measure the structure and function of the brain. The results being reported apply only to Aim 4 of the grant.
Period: Overall Study
Arm/Group | Alcohol Group | No Alcohol Group
Started | 5 | 4
Completed | 5 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Alcohol Group: Participants who have recently consumed alcohol.
  MRI Scanner: Participants will enter the MRI scanner and complete a series of computer tasks that include noise blasts while undergoing brain scans that measure the structure and function of the brain. We are reporting the data per sequence. The results being reported apply only to Aim 4 of the grant.
  The results being reported apply only to Aim 4 of the grant. Aims 1-3 focused on analyzing existing archival genomic data and were covered by another protocol, which was not entered into CT.gov, as those aims did not meet the definition of a clinical trial and were approved under a different IRB protocol number and approval process than Aim 4. All participants only completed one session, but within that one session, they completed the loud noises task two times in a row on the same MRI scan, it was done twice to get a more reliable answer when the two measures were combined.
- No Alcohol Group: Participants who have not recently consumed alcohol.
  MRI Scanner: Participants will enter the MRI scanner and complete a series of computer tasks that include noise blasts while undergoing brain scans that measure the structure and function of the brain. We are reporting the data per sequence. The results being reported apply only to Aim 4 of the grant.
  The results being reported apply only to Aim 4 of the grant. Aims 1-3 focused on analyzing existing archival genomic data and were covered by another protocol, which was not entered into CT.gov, as those aims did not meet the definition of a clinical trial and were approved under a different IRB protocol number and approval process than Aim 4. All participants only completed one session, but within that one session, they completed the loud noises task two times in a row on the same MRI scan, it was done twice to get a more reliable answer when the two measures were combined.
- Total: Total of all reporting groups
Arm/Group | Alcohol Group | No Alcohol Group | Total
Number analyzed (Participants) | 5 | 4 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 4 | 9
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.2 (6.8) | 27.75 (5.74) | 27.96 (6.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 3 | 3 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 4 | 2 | 6
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Changes in Alcohol-influenced Behavior
Description: Aggressive behavior (i.e., the average volume of noise blasts selected to be administered to participants' opponents) after recent consumption of an alcoholic beverages (versus without recent consumption of an alcoholic beverages) will be measured using the validated and computerized Taylor Competitive Reaction-Time Task. The Taylor Competitive Reaction-Time Task consists of multiple trials that each assess aggression, via a four-point scale that ranges from 1 (low noise blast volume [low aggression]) to 4 (high noise blast volume [high aggression]). Noise blast settings are averaged to provide a total score ranging from 1 to 4, with higher scores indicating greater aggression.
Time Frame: During the course of the MRI session
Population: The results apply only to Aim 4. Aims 1-3 were covered by another protocol that did not meet the definition of a ct and were approved under a different IRB protocol #. All participants completed only one session, but within that session, they performed the loud noises task twice consecutively on the same MRI scan.It was done twice to get a more reliable answer when the two measures were combined.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Alcohol Group: Participants who have recently consumed alcohol.
  MRI Scanner: Participants will enter the MRI scanner and complete a series of computer tasks that include noise blasts while undergoing brain scans that measure the structure and function of the brain.
  We are reporting the data per sequence. The results being reported apply only to Aim 4 of the grant. Aims 1-3 focused on analyzing existing archival genomic data. Aim 4 is the only one that met the definition of clinical trial. Aims 1-3 were covered by another protocol, that was not entered into CT.gov since it did not meet the definition of a clinical trial.
- No Alcohol Group: Participants who have not recently consumed alcohol.
  MRI Scanner: Participants will enter the MRI scanner and complete a series of computer tasks that include noise blasts while undergoing brain scans that measure the structure and function of the brain. Aims 1-3 were covered by another protocol, that was not entered into CT.gov since it did not meet the definition of a clinical trial.
  We are reporting the data per sequence. The results being reported apply only to Aim 4 of the grant. Aims 1-3 focused on analyzing existing archival genomic data. Aim 4 is the only one that met the definition of clinical trial..
Arm/Group | Alcohol Group | No Alcohol Group
Number analyzed (Participants) | 5 | 4
units on a scale | 1.56 (.72) | 1.49 (.56)

ADVERSE EVENTS:
Time Frame: Duration of the one-day session, including the MRI scan and the computer tasks. The data was only collected during the one-day session.
Description: Self-report by the participants
Groups:
- Alcohol Group: Participants who have recently consumed alcohol.
  MRI Scanner: Participants will enter the MRI scanner and complete a series of computer tasks that include noise blasts while undergoing brain scans that measure the structure and function of the brain
  The results being reported apply only to Aim 4 of the grant. Aims 1-3 focused on analyzing existing archival genomic data and were covered by another protocol, which was not entered into CT.gov, as those aims did not meet the definition of a clinical trial and were approved under a different IRB protocol number and approval process than Aim 4. All participants only completed one session, but within that one session, they completed the loud noises task two times in a row on the same MRI scan, it was done twice to get a more reliable answer when the two measures were combined.
- No Alcohol Group: Participants who have not recently consumed alcohol.
  MRI Scanner: Participants will enter the MRI scanner and complete a series of computer tasks that include noise blasts while undergoing brain scans that measure the structure and function of the brain
  The results being reported apply only to Aim 4 of the grant. Aims 1-3 focused on analyzing existing archival genomic data and were covered by another protocol, which was not entered into CT.gov, as those aims did not meet the definition of a clinical trial and were approved under a different IRB protocol number and approval process than Aim 4. All participants only completed one session, but within that one session, they completed the loud noises task two times in a row on the same MRI scan, it was done twice to get a more reliable answer when the two measures were combined.
Arm/Group | Alcohol Group | No Alcohol Group
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/4
Other Adverse Events (participants affected / at risk) | 0/5 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-08-24): https://cdn.clinicaltrials.gov/large-docs/45/NCT03725345/Prot_SAP_001.pdf
  • Informed Consent Form (2022-09-27): https://cdn.clinicaltrials.gov/large-docs/45/NCT03725345/ICF_000.pdf